CLINICAL TRIAL: NCT00261612
Title: Bortezomib, Rituximab and Dexamethasone (BORID) for Relapsed/Refractory Mantle Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-002150-64; MCL 03
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2006-10-18 (Estimated); Status verified 2006-10

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: relapsed or chemotherapy-refractory disease
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — Bortezomib; Rituximab; Dexamethasone; Clinical Protocols

INTERVENTIONS:
Drug: bortezomib
Drug: rituximab
Drug: dexamethasone
Procedure: treatment protocol

SUMMARY:
Mantle cell lymphoma (MCL) remains difficult to treat by standard treatment approaches. Novel drugs have shown promising results in early clinical evaluations. In the current trial, we investigate a combination of bortezomib (a proteasome inhibitor), rituximab (a monoclonal antibody), and dexamethasone in patients with MCL, who have already been pretreated by standard chemotherapy and show again signs of disease progression. The study objectives include remission rates, safety of this drug combination, and survival time.

DETAILED DESCRIPTION:
Description of the treatment regimen: Bortezomib: 1.3 mg/m2 as i.v. bolus injection, given on days 1, 4, 8, and 11 of each treatment cycle; Rituximab: 375 mg/m2 infusion, day 1 of each cycle; Dexamethasone: 40 mg per day orally (days 1 - 4) of each treatment cycle. Treatment will be given for a total of 6 cycles (every 21 days), followed by maintenance treatment with rituximab (375 mg/m2 every two months for 4 times)

ELIGIBILITY:
Inclusion Criteria:

* mantle cell lymphoma at stage II - IV, previously treated with at least one line of prior therapy (CHOP or CHOP-like), measurable disease, age 19 - 75 years, adequate cardiac, liver and renal function tests, patient's written informed consent

Exclusion Criteria:

* second malignancy, evidence for CNS involvement, clinically significant peripheral neuropathy (grade II or higher), HIV positivity, pregnancy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2005-01; Study Completion 2007-01

PRIMARY OUTCOMES:
response rate

SECONDARY OUTCOMES:
safety
progression free survival
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Drach, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Medical University Vienna, Dept. of Medicine I, Clinical Division of Oncology, Vienna, Austria

REFERENCES:
- [Background] Drach J, Seidl S, Kaufmann H. Treatment of mantle cell lymphoma: targeting the microenvironment. Expert Rev Anticancer Ther. 2005 Jun;5(3):477-85. doi: 10.1586/14737140.5.3.477. PMID 16001955
- [Background] Kaufmann H, Raderer M, Wohrer S, Puspok A, Bankier A, Zielinski C, Chott A, Drach J. Antitumor activity of rituximab plus thalidomide in patients with relapsed/refractory mantle cell lymphoma. Blood. 2004 Oct 15;104(8):2269-71. doi: 10.1182/blood-2004-03-1091. Epub 2004 May 27. PMID 15166030
- [Derived] Lamm W, Kaufmann H, Raderer M, Hoffmann M, Chott A, Zielinski C, Drach J. Bortezomib combined with rituximab and dexamethasone is an active regimen for patients with relapsed and chemotherapy-refractory mantle cell lymphoma. Haematologica. 2011 Jul;96(7):1008-14. doi: 10.3324/haematol.2011.041392. Epub 2011 Apr 12. PMID 21486866